CLINICAL TRIAL: NCT03985046
Title: A Pilot Study of Sintilimab Plus Chemotherapy Followed by Definitive Concurrent Chemoradiotherapy in Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Sintilimab Plus Chemotherapy Followed by dCRT in Locally Advanced ESCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Kuai Le Zhao, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESO-Shanghai14
Record Dates: First submitted 2019-06-10; First posted 2019-06-13 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab plus chemotherapy (Experimental)
  Interventions: Drug: Sintilimab plus Chemotherapy

INTERVENTIONS:
Drug: Sintilimab plus Chemotherapy — Sintilimab will be administered intravenously, a fixed dose of 200 mg. Paclitaxel 135mg/m2, carboplatin AUC=5. Once every 3 weeks.

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of A sintilimab plus chemotherapy followed by definitive concurrent chemoradiotherapy in locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Aged 18-75 years
3. Histologically confirmed esophageal squamous cell carcinoma
4. Clinical stages T3-4N0M0 or TxN1M0 or TxNxM1a or TxNxM1b (Only for cervical lymph nodes or celiac lymph nodes metastasis) based on the 6th UICC-TNM classification

7. Eastern Cooperative Oncology Group(ECOG) performance status: 0-1 8. Life expectancy ≥3 months 9. Adequate organ functions Absolute neutrophil counts (ANC) ≥1.5×109⁄L; Hemoglobin (Hb) ≥9g⁄dl; Platelet (Plt) ≥100×109⁄L; Total bilirubin ≤1.5 upper limit of normal (ULN); Aspartate transaminase (AST) ≤2.5 ULN; Alanine aminotransferase (ALT) ≤2.5 ULN; Creatinine ≤1.5 ULN

Exclusion Criteria:

1. Esophageal perforation or hematemesis
2. Any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism and hypothyroidism (effective hormone replacement therapy excepted)) and immunosuppressive agents or systemic hormonal therapy indicated within 28 days (for adverse events of chemoradiotherapy excepted).
3. Previously received or receiving other PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1.
4. Allergic to macromolecular protein preparations, or to any of the ingredients in sintilimab for injection.
5. Uncontrolled heart diseases or clinical symptoms, such as: (1) New York Heart Association(NYHA) class II or higher heart failure; (2) unstable angina; (3) myocardial infarction within 1 year; (4)clinically significant arrhythmia requiring clinical intervention.
6. Congenital or acquired immunodeficiency (such as HIV infection); active hepatitis B (HBV-DNA≥104 copy number/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the detection limit of the analytical method); active tuberculosis.
7. Active infection or unexplained fever >38.5 °C within 2 weeks before randomization (fever due to tumor excepted, according to investigator).
8. Patients with fertility reluctant to take contraceptive measures during the trial, or female patients pregnant or breastfeeding.
9. According to the investigator, other factors that may cause termination of the study. ie, other serious diseases (including mental illness) require combined treatment, family or social factors, which may affect the safety or the collection of trial data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Local Control Rate | up to 42 months

SECONDARY OUTCOMES:
Adverse Events | up to 42 months
Progression-free Survival | up to 42 months
Overall Survival | up to 42 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ai D, Hao S, Shen W, Wu Q, Zhang S, Chen Y, Liu Q, Deng J, Zhu H, Chen K, Mo M, Gu D, Liu Y, Zhang Z, Zhou G, Hu J, Zhang Z, Ye J, Zhao K. Induction sintilimab and chemotherapy followed by concurrent chemoradiotherapy for locally advanced esophageal cancer: a proof-of-concept, single-arm, multicenter, phase 2 trial. EClinicalMedicine. 2024 Feb 6;69:102471. doi: 10.1016/j.eclinm.2024.102471. eCollection 2024 Mar. PMID 38356729